CLINICAL TRIAL: NCT04432623
Title: A Phase 1b Sequential Open Label Dose-Ranging Study of Safety, Pharmacokinetics, and Preliminary Activity of Benserazide in Subjects With Beta Thalassemia Intermedia and Sickle Cell Disease
Brief Title: The BENeFiTS Trial in Beta Thalassemia Intermedia
Acronym: PB04-001
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Phoenicia BioScience (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB04-001; R33HL147845 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Beta Thalassemia Intermedia; Sickle Cell Disease
Keywords: Non-transfusion dependent beta thalassemia; Sickle cell disease
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Each higher dose level cohort will be enrolled after 2 weeks of treatment in the lower dose level. Additional doses or regimens may be added or expanded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Low dose (Experimental): A low dose, by mouth, once per day, on Monday, Wednesday, and Friday for 12 weeks
  Interventions: Drug: Benserazide Only Product
- Middle dose (Experimental): A middle dose, by mouth, once per day, on Monday, Wednesday, and Friday, for 12 weeks
  Interventions: Drug: Benserazide Only Product
- High dose 3 days per week (Experimental): Highest dose, by mouth, once per day, on Monday, Wednesday, and Friday, for 12 to 24 weeks
  Interventions: Drug: Benserazide Only Product
- High dose 5 days per week (Experimental): The highest dose, by mouth once per day on 5 days per week for 24 weeks
  Interventions: Drug: Benserazide Only Product
- Sickle Cell Disease Arm (Experimental): The most active dose given once per day on the most active regimen for up 24 weeks
  Interventions: Drug: Benserazide Only Product

INTERVENTIONS:
Drug: Benserazide Only Product — Investigational drug

SUMMARY:
Beta-thalassemias and hemoglobinopathies are serious inherited blood diseases caused by abnormal or deficiency of beta A chains of hemoglobin, the protein in red blood cells which delivers oxygen throughout the body.The diseases are characterized by hemolytic anemia, organ damage, and early mortality without treatment. Increases in another type of (normal) hemoglobin, fetal globin (HbF), which is normally silenced in infancy, reduces anemia and morbidity. Even incremental augmentation of fetal globin is established to reduce red blood cell pathology, anemia, certain complications, and to improve survival.

This trial will evaluate an oral drug discovered in a high throughput screen, which increases fetal globin protein (HbF and red blood cells expressing HbF)and messenger ribonucleic acid (mRNA) to high levels in anemic nonhuman primates and in transgenic mice. The study drug acts by suppressing 4 repressors of the fetal globin gene promoter in progenitor cells from patients. The drug has been used for 50 years in a combination product for different actions - to enhance half-life and reduce side effects of a different active drug- and is considered safe for long-term use.

This trial will first evaluate 3 dose levels in small cohorts of nontransfused patients with beta thalassemia intermedia. The most active dose will then be evaluated in larger subject groups with beta thalassemia and other hemoglobinopathies, such as sickle cell disease.

DETAILED DESCRIPTION:
The study will first evaluate 3 doses of the investigational drug which are considered safe with chronic use in a combination therapeutic used widely for a different disease in Europe and Canada. The doses to be studied are human equivalent doses of doses that are active in nonhuman primates in inducing high level fetal globin messenger ribonucleic acid (mRNA), protein, and proportions of red blood cells expressing fetal globin protein (F-cells). Additive effects are observed with hydroxyurea in sickle cell patients' cells in vitro.

The study will first evaluate the study therapeutic in male and female patients who are 18 years and older. After a screening period to obtain baseline medical and laboratory data, the study drug will be taken by mouth once per day, every other day. The first dose will be taken in a clinical unit, and thereafter will be taken at home for 12 weeks. Laboratory tests, physical exams, and tolerability will be assessed 6 times over 4 months, including for one month after completion of dosing.

The cohorts will be enrolled sequentially. Each new cohort will begin after the prior lower dose cohort has received 2 weeks of treatment without serious adverse events related to the study drug. The dose that increases fetal globin assays to the highest degree will be evaluated in a larger group of subjects with beta thalassemia intermedia and a groups with sickle cell disease. Other regimens or test doses may be added as needed to identify an active dose and regimen. The study drug is expected to be safe when added to most other medications used to treat thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia intermedia (BTI) or (NTDT, Non-Transfusion Dependent Thalassemia) with at least one documented beta thalassemia mutation, including HbE beta thalassemia or an established diagnosis of sickle cell disease
* >18 years of age at time of consent
* Average of 2 total hemoglobin (Hgb) levels between 6.0 and 10.0 g/dL in the preceding 6 months
* Able and willing to give consent and comply with all study procedures
* If female and of childbearing potential, must have a documented negative pregnancy test prior to entry and agree to use one or more locally medically accepted methods of contraception

Exclusion Criteria:

* Red blood cell (RBC) transfusion within 2 months prior to administration of study medication
* Participating in a chronic transfusion program
* Pulmonary hypertension requiring oxygen therapy
* Use of erythropoiesis stimulating agents within 90 days of first dose
* Transaminases > 3 times upper limit of institution normal (ULN)
* Total and direct bilirubin > 3 times institution ULN unless due solely to hemolysis
* Known infection with HIV or hepatitis C (untreated)
* Fever > 38.5°C in the week prior to first administration of study medication
* History of osteoporosis or osteomalacia with a fragility fracture
* Received other investigational systemic therapy within 30 days prior to first dose
* Narrow angle glaucoma
* Currently pregnant or breast feeding a child
* Known current drug or alcohol abuse
* Taking monoamine oxidase inhibitors
* Other co-morbidity that substantially increases subject risk for the study per Investigator discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 12 to 24 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Maximum plasma concentration (Cmax) | 4 weeks
  drug concentration (ng/ml)
Plasma drug concentration over time | 4 weeks
  Area under the curve

SECONDARY OUTCOMES:
F-cells | 12 to 24 weeks
  % Red blood cells containing HbF
HbF protein per cell | 12 to 24 weeks
  Mean fluorescent intensity (MFI)
Fetal hemoglobin (HbF) | 12 to 24 weeks
  % and absolute (g/dl)
Hemoglobin | 16 to 24 weeks
  gram/dl

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perrine, MD, Study Director — Phoenicia BioScience; Kevin Kuo, MD, Principal Investigator — University Health Network, Toronto General Hospital; Sylvia Singer, MD, Principal Investigator — UCSF Benioff Children's Hospital at Oakland; Hanny D Al-Samkari, MD, Principal Investigator — Massachusetts General Hospital; Sujit Sheth, MD MS, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (4):
  - UCSF Benioff Children's Hospital at Oakland, Oakland, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Susan Perrine, Weston, Massachusetts
  - Weil Cornell Medicine, New York, New York
- University Health Network and Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Results will be provided in abstracts as the study is being conducted and in a publication after completion and analysis.

REFERENCES:
- [Background] Boosalis MS, Sangerman JI, White GL, Wolf RF, Shen L, Dai Y, White E, Makala LH, Li B, Pace BS, Nouraie M, Faller DV, Perrine SP. Novel Inducers of Fetal Globin Identified through High Throughput Screening (HTS) Are Active In Vivo in Anemic Baboons and Transgenic Mice. PLoS One. 2015 Dec 29;10(12):e0144660. doi: 10.1371/journal.pone.0144660. eCollection 2015. PMID 26713848
- [Background] Dai Y, Sangerman J, Luo HY, Fucharoen S, Chui DH, Faller DV, Perrine SP. Therapeutic fetal-globin inducers reduce transcriptional repression in hemoglobinopathy erythroid progenitors through distinct mechanisms. Blood Cells Mol Dis. 2016 Jan;56(1):62-9. doi: 10.1016/j.bcmd.2015.10.004. Epub 2015 Oct 27. PMID 26603726
- [Background] Dai Y, Sangerman J, Nouraie M, Faller AD, Oneal P, Rock A, Owoyemi O, Niu X, Nekhai S, Maharaj D, Cui S, Taylor R, Steinberg M, Perrine S. Effects of hydroxyurea on F-cells in sickle cell disease and potential impact of a second fetal globin inducer. Am J Hematol. 2017 Jan;92(1):E10-E11. doi: 10.1002/ajh.24590. Epub 2016 Nov 18. No abstract available. PMID 27766663
- [Background] Chen Z, Luo HY, Steinberg MH, Chui DH. BCL11A represses HBG transcription in K562 cells. Blood Cells Mol Dis. 2009 Mar-Apr;42(2):144-9. doi: 10.1016/j.bcmd.2008.12.003. Epub 2009 Jan 18. PMID 19153051
- [Background] Sedgewick AE, Timofeev N, Sebastiani P, So JCC, Ma ESK, Chan LC, Fucharoen G, Fucharoen S, Barbosa CG, Vardarajan BN, Farrer LA, Baldwin CT, Steinberg MH, Chui DHK. BCL11A is a major HbF quantitative trait locus in three different populations with beta-hemoglobinopathies. Blood Cells Mol Dis. 2008 Nov-Dec;41(3):255-258. doi: 10.1016/j.bcmd.2008.06.007. Epub 2008 Aug 8. PMID 18691915
- [Background] Zhou D, Liu K, Sun CW, Pawlik KM, Townes TM. KLF1 regulates BCL11A expression and gamma- to beta-globin gene switching. Nat Genet. 2010 Sep;42(9):742-4. doi: 10.1038/ng.637. Epub 2010 Aug 1. PMID 20676097
- [Background] Cao H, Stamatoyannopoulos G, Jung M. Induction of human gamma globin gene expression by histone deacetylase inhibitors. Blood. 2004 Jan 15;103(2):701-9. doi: 10.1182/blood-2003-02-0478. Epub 2003 Aug 14. PMID 12920038
- [Background] Franco RS, Yasin Z, Palascak MB, Ciraolo P, Joiner CH, Rucknagel DL. The effect of fetal hemoglobin on the survival characteristics of sickle cells. Blood. 2006 Aug 1;108(3):1073-6. doi: 10.1182/blood-2005-09-008318. PMID 16861353
- [Background] Perrine RP, Brown MJ, Clegg JB, Weatherall DJ, May A. Benign sickle-cell anaemia. Lancet. 1972 Dec 2;2(7788):1163-7. doi: 10.1016/s0140-6736(72)92592-5. No abstract available. PMID 4117591
- [Background] Wang X, Thein SL. Switching from fetal to adult hemoglobin. Nat Genet. 2018 Apr;50(4):478-480. doi: 10.1038/s41588-018-0094-z. PMID 29610477
- [Background] Singer ST, Kuypers FA, Olivieri NF, Weatherall DJ, Mignacca R, Coates TD, Davies S, Sweeters N, Vichinsky EP; E/beta Thalassaemia Study Group. Fetal haemoglobin augmentation in E/beta(0) thalassaemia: clinical and haematological outcome. Br J Haematol. 2005 Nov;131(3):378-88. doi: 10.1111/j.1365-2141.2005.05768.x. PMID 16225658
- [Background] Perrine SP, Mankidy R, Boosalis MS, Bieker JJ, Faller DV. Erythroid Kruppel-like factor (EKLF) is recruited to the gamma-globin gene promoter as a co-activator and is required for gamma-globin gene induction by short-chain fatty acid derivatives. Eur J Haematol. 2009 Jun;82(6):466-76. doi: 10.1111/j.1600-0609.2009.01234.x. Epub 2009 Feb 5. PMID 19220418
- [Background] Tanabe O, McPhee D, Kobayashi S, Shen Y, Brandt W, Jiang X, Campbell AD, Chen YT, Chang Cs, Yamamoto M, Tanimoto K, Engel JD. Embryonic and fetal beta-globin gene repression by the orphan nuclear receptors, TR2 and TR4. EMBO J. 2007 May 2;26(9):2295-306. doi: 10.1038/sj.emboj.7601676. Epub 2007 Apr 12. PMID 17431400
- [Background] Borg J, Papadopoulos P, Georgitsi M, Gutierrez L, Grech G, Fanis P, Phylactides M, Verkerk AJ, van der Spek PJ, Scerri CA, Cassar W, Galdies R, van Ijcken W, Ozgur Z, Gillemans N, Hou J, Bugeja M, Grosveld FG, von Lindern M, Felice AE, Patrinos GP, Philipsen S. Haploinsufficiency for the erythroid transcription factor KLF1 causes hereditary persistence of fetal hemoglobin. Nat Genet. 2010 Sep;42(9):801-5. doi: 10.1038/ng.630. Epub 2010 Aug 1. PMID 20676099
- [Background] Atweh GF, Sutton M, Nassif I, Boosalis V, Dover GJ, Wallenstein S, Wright E, McMahon L, Stamatoyannopoulos G, Faller DV, Perrine SP. Sustained induction of fetal hemoglobin by pulse butyrate therapy in sickle cell disease. Blood. 1999 Mar 15;93(6):1790-7. PMID 10068649
- [Background] Centis F, Tabellini L, Lucarelli G, Buffi O, Tonucci P, Persini B, Annibali M, Emiliani R, Iliescu A, Rapa S, Rossi R, Ma L, Angelucci E, Schrier SL. The importance of erythroid expansion in determining the extent of apoptosis in erythroid precursors in patients with beta-thalassemia major. Blood. 2000 Nov 15;96(10):3624-9. PMID 11071663
- [Background] Collins AF, Pearson HA, Giardina P, McDonagh KT, Brusilow SW, Dover GJ. Oral sodium phenylbutyrate therapy in homozygous beta thalassemia: a clinical trial. Blood. 1995 Jan 1;85(1):43-9. PMID 7528572
- [Background] Niihara Y, Miller ST, Kanter J, Lanzkron S, Smith WR, Hsu LL, Gordeuk VR, Viswanathan K, Sarnaik S, Osunkwo I, Guillaume E, Sadanandan S, Sieger L, Lasky JL, Panosyan EH, Blake OA, New TN, Bellevue R, Tran LT, Razon RL, Stark CW, Neumayr LD, Vichinsky EP; Investigators of the Phase 3 Trial of l-Glutamine in Sickle Cell Disease. A Phase 3 Trial of l-Glutamine in Sickle Cell Disease. N Engl J Med. 2018 Jul 19;379(3):226-235. doi: 10.1056/NEJMoa1715971. PMID 30021096
- [Background] Minniti CP. l-Glutamine and the Dawn of Combination Therapy for Sickle Cell Disease. N Engl J Med. 2018 Jul 19;379(3):292-294. doi: 10.1056/NEJMe1800976. No abstract available. PMID 30021091
- [Background] Kato GJ, Gladwin MT, Steinberg MH. Deconstructing sickle cell disease: reappraisal of the role of hemolysis in the development of clinical subphenotypes. Blood Rev. 2007 Jan;21(1):37-47. doi: 10.1016/j.blre.2006.07.001. Epub 2006 Nov 7. PMID 17084951
- [Background] Saraf S, Farooqui M, Infusino G, Oza B, Sidhwani S, Gowhari M, Vara S, Gao W, Krauz L, Lavelle D, DeSimone J, Molokie R, Saunthararajah Y. Standard clinical practice underestimates the role and significance of erythropoietin deficiency in sickle cell disease. Br J Haematol. 2011 May;153(3):386-92. doi: 10.1111/j.1365-2141.2010.08479.x. Epub 2011 Mar 21. PMID 21418176
- [Background] Perrine SP, Pace BS, Faller DV. Targeted fetal hemoglobin induction for treatment of beta hemoglobinopathies. Hematol Oncol Clin North Am. 2014 Apr;28(2):233-48. doi: 10.1016/j.hoc.2013.11.009. PMID 24589264
- [Background] Steinberg MH, Rodgers GP. Pharmacologic modulation of fetal hemoglobin. Medicine (Baltimore). 2001 Sep;80(5):328-44. doi: 10.1097/00005792-200109000-00007. No abstract available. PMID 11552087
- [Background] Weatherall DJ. The inherited diseases of hemoglobin are an emerging global health burden. Blood. 2010 Jun 3;115(22):4331-6. doi: 10.1182/blood-2010-01-251348. Epub 2010 Mar 16. PMID 20233970
- [Background] Taher AT, Cappellini MD. How I manage medical complications of beta-thalassemia in adults. Blood. 2018 Oct 25;132(17):1781-1791. doi: 10.1182/blood-2018-06-818187. Epub 2018 Sep 11. PMID 30206117
- [Background] Borgna-Pignatti C. Modern treatment of thalassaemia intermedia. Br J Haematol. 2007 Aug;138(3):291-304. doi: 10.1111/j.1365-2141.2007.06654.x. Epub 2007 Jun 12. PMID 17565568
- [Background] Sripichai O, Makarasara W, Munkongdee T, Kumkhaek C, Nuchprayoon I, Chuansumrit A, Chuncharunee S, Chantrakoon N, Boonmongkol P, Winichagoon P, Fucharoen S. A scoring system for the classification of beta-thalassemia/Hb E disease severity. Am J Hematol. 2008 Jun;83(6):482-4. doi: 10.1002/ajh.21130. PMID 18186524
- [Background] Nuinoon M, Makarasara W, Mushiroda T, Setianingsih I, Wahidiyat PA, Sripichai O, Kumasaka N, Takahashi A, Svasti S, Munkongdee T, Mahasirimongkol S, Peerapittayamongkol C, Viprakasit V, Kamatani N, Winichagoon P, Kubo M, Nakamura Y, Fucharoen S. A genome-wide association identified the common genetic variants influence disease severity in beta0-thalassemia/hemoglobin E. Hum Genet. 2010 Mar;127(3):303-14. doi: 10.1007/s00439-009-0770-2. PMID 20183929
- [Background] Uda M, Galanello R, Sanna S, Lettre G, Sankaran VG, Chen W, Usala G, Busonero F, Maschio A, Albai G, Piras MG, Sestu N, Lai S, Dei M, Mulas A, Crisponi L, Naitza S, Asunis I, Deiana M, Nagaraja R, Perseu L, Satta S, Cipollina MD, Sollaino C, Moi P, Hirschhorn JN, Orkin SH, Abecasis GR, Schlessinger D, Cao A. Genome-wide association study shows BCL11A associated with persistent fetal hemoglobin and amelioration of the phenotype of beta-thalassemia. Proc Natl Acad Sci U S A. 2008 Feb 5;105(5):1620-5. doi: 10.1073/pnas.0711566105. Epub 2008 Feb 1. PMID 18245381
- [Background] Labie D, Pagnier J, Lapoumeroulie C, Rouabhi F, Dunda-Belkhodja O, Chardin P, Beldjord C, Wajcman H, Fabry ME, Nagel RL. Common haplotype dependency of high G gamma-globin gene expression and high Hb F levels in beta-thalassemia and sickle cell anemia patients. Proc Natl Acad Sci U S A. 1985 Apr;82(7):2111-4. doi: 10.1073/pnas.82.7.2111. PMID 2580306
- [Background] Silva M, Grillot D, Benito A, Richard C, Nunez G, Fernandez-Luna JL. Erythropoietin can promote erythroid progenitor survival by repressing apoptosis through Bcl-XL and Bcl-2. Blood. 1996 Sep 1;88(5):1576-82. PMID 8781412
- [Background] Pootrakul P, Sirankapracha P, Hemsorach S, Moungsub W, Kumbunlue R, Piangitjagum A, Wasi P, Ma L, Schrier SL. A correlation of erythrokinetics, ineffective erythropoiesis, and erythroid precursor apoptosis in thai patients with thalassemia. Blood. 2000 Oct 1;96(7):2606-12. PMID 11001918
- [Background] Singer ST, Vichinsky EP, Sweeters N, Rachmilewitz E. Darbepoetin alfa for the treatment of anaemia in alpha- or beta- thalassaemia intermedia syndromes. Br J Haematol. 2011 Jul;154(2):281-4. doi: 10.1111/j.1365-2141.2011.08617.x. Epub 2011 Apr 18. No abstract available. PMID 21496003